CLINICAL TRIAL: NCT04946903
Title: A Randomized, Open Label, Single Dose, 2-way Crossover Clinical Trial to Evaluate the Pharmacokinetic Characteristics and Safety Between HCP1902 and RLD2007/RLD2008 in Healthy Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety Between HCP1902 and Co-administration of RLD2007, RLD2008
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-DATA-101
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Period 1: Fasted state + RLD2007 +RLD2008,
  Period 2: Fasted state + HCP1902
  Interventions: Drug: RLD2007; Drug: RLD2008; Drug: HCP1902
- Sequence 2 (Experimental): Period 1: Fasted state + HCP1902,
  Period 2: Fasted state + RLD2007 + RLD2008
  Interventions: Drug: RLD2007; Drug: RLD2008; Drug: HCP1902

INTERVENTIONS:
Drug: RLD2007 — Take it once per period.
Drug: RLD2008 — Take it once per period.
Drug: HCP1902 — Take it once per period.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic characteristics and safety between HCP1902 and co-administration of RLD2007/RLD2008 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Age 19~54 years in healthy volunteers 19 kg/m^2 ≤ BMI < 28 kg/m^2, weight(men) ≥55kg / weight(women) ≥45kg
* 90 mmHg ≤ SBP <140 mmHg, 50 mmHg ≤ DBP <90 mmHg
* agrees that the person, spouse, or partner uses appropriate medically recognized contraception and does not provide sperm or eggs from the date of administration of the first investigational drug to 7 days after the administration of the last investigational drug.
* Subjects who voluntarily decides to participate in this clinical trial and agree in writing to ensure compliance with the clinical trial

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
* Subjects who judged ineligible by the investigator

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
AUCt | 0~48 hour
  Pharmacokinetic evaluation
Cmax | 0~48 hour
  Pharmacokinetic evaluation

SECONDARY OUTCOMES:
AUCinf | 0~48 hour
  Pharmacokinetic evaluation
Tmax | 0~48 hour
  Pharmacokinetic evaluation
t1/2 | 0~48 hour
  Pharmacokinetic evaluation
CL/F | 0~48 hour
  Pharmacokinetic evaluation
Vd/F | 0~48 hour
  Pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Mingeul Kim, Principal Investigator — Jeonbuk University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea